CLINICAL TRIAL: NCT00118508
Title: The Prevention of Osteoporosis in Premenopausal and Newly Postmenopausal (Up to 8 Years) Women With Breast Cancer Following Chemotherapy (REBBeCA Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Procter and Gamble (Industry); Aventis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Susan L. Greenspan, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB#0404173
Record Dates: First submitted 2005-06-30; First posted 2005-07-11 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Placebo Comparator): Group A will receive active study drug
  Interventions: Drug: risedronate (including placebo)

INTERVENTIONS:
Drug: risedronate (including placebo) — risedronate 35mg weekly
  Other Names: Actonel

SUMMARY:
The purpose of this study is to evaluate the effectiveness of once weekly risedronate in the prevention and treatment of bone loss in premenopausal and newly menopausal women with breast cancer who have received chemotherapy.

The hypothesis is that bisphosphonate therapy will prevent bone loss at clinically relevant sites, such as the hip and spine. The investigators also hypothesize that there will be a correlation between biochemical markers of bone turnover and changes in bone mineral density.

DETAILED DESCRIPTION:
Breast cancer is a significant public health problem accounting for approximately 30% of new cancers diagnosed annually. Much advancement has been made in the treatment of these cancers which has significantly decreased the mortality rates. Treatment, including adjuvant chemotherapy and hormonal therapy, prolongs disease free survival and overall survival of patients with breast cancer. The cytotoxic drugs, however, can cause premature ovarian failure and subsequent menopause. This risk has been reported to range from 53% to 89%. Temporary or permanent chemotherapy induced ovarian failure is important because of potential bone loss associated with the estrogen loss. Initiating a potent antiresorptive agent, risedronate, should prevent or improve bone mass in these women.

Comparison: The investigators will compare bone mass/markers of study subjects receiving risedronate with study subjects receiving placebo. All subjects will be provided calcium and vitamin D supplementation as needed.

ELIGIBILITY:
Inclusion Criteria:

* Pre- and newly postmenopausal (up to 8 years) women ages 18 and older
* Breast cancer treated with chemotherapeutic agents, with or without tamoxifen/aromatase inhibitors
* Negative pregnancy test

Exclusion Criteria:

* Stage 4 breast cancer
* Any illness or medications known to affect bone metabolism
* History of osteoporosis or history of vertebral or hip fractures
* Kidney stones in the past 5 years
* Active peptic ulcer disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2003-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
That bone loss, as determined through BMD every six months, will be prevented at clinically relevant sites, such as the hip & spine, through the use of bisphosphonate therapy in study subjects. | 24 months

SECONDARY OUTCOMES:
There will be a correlation between biochemical markers of bone turnover and changes in BMD. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Greenspan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center (GCRC), Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Greenspan SL, Brufsky A, Lembersky BC, Bhattacharya R, Vujevich KT, Perera S, Sereika SM, Vogel VG. Risedronate prevents bone loss in breast cancer survivors: a 2-year, randomized, double-blind, placebo-controlled clinical trial. J Clin Oncol. 2008 Jun 1;26(16):2644-52. doi: 10.1200/JCO.2007.15.2967. Epub 2008 Apr 21. PMID 18427147